CLINICAL TRIAL: NCT04802304
Title: Beyond Bias - Reducing Provider Bias Towards Adolescents to Increase Contraception Take-Up in Tanzania, Burkina Faso, and Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of California, Los Angeles (Other); Bill and Melinda Gates Foundation (Other); Pathfinder International (Industry)
Responsible Party: Principal Investigator, Zachary Wagner, Professor of Policy Analysis, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0387
Record Dates: First submitted 2021-01-29; First posted 2021-03-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Family Planning Services
Keywords: Human-centered design; Health provider bias

STUDY DESIGN:
Intervention Model Description: Half of the eligible clinics in each country (233 in total) are randomly assigned to receive the intervention, while the remaining half serves as control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Beyond Bias Treatment
- Control (No Intervention)

INTERVENTIONS:
Other: Beyond Bias Treatment — The intervention has three components: 1) a summit that includes impactful stories told to and by family planning providers that highlight the consequences of provider bias, 2) a forum for continued communication between providers, and 3) a rewards program where clinics in which providers exhibit less biased client interactions or who have improved the most towards this end will be rewarded with social recognition and a ceremony.
  Arms: Treatment

SUMMARY:
Beyond Bias will evaluate the impact of an intervention designed to reduce family planning provider bias towards young, unmarried, and nulliparous women in Tanzania, Burkina Faso, and Pakistan. The intervention has three components: 1) a summit that includes impactful stories told to and by family planning providers that highlight the consequences of provider bias, 2) a forum for continued communication between providers, and 3) a rewards program where clinics in which providers exhibit less biased client interactions or who have improved the most towards this end will be rewarded with social recognition and a ceremony.

Half of the eligible clinics in each country (233 in total) are randomly assigned to receive the intervention, while the remaining half serves as control. The objective of the evaluation is to estimate the impact of the intervention on a range of outcomes related to quality of family planning care among young, unmarried, and nulliparous women. The investigators hypothesize that the intervention will increase the share of young, unmarried, and nulliparous women who received counseling on a range of methods, counseling on long acting methods, and who received their preferred method.

The investigators will collect four types of data to evaluate the intervention: 1) provider surveys, 2) mystery clients' visits, 3) direct observations of client-provider interactions, and 4) qualitative interviews with clients, providers, and implementors.

ELIGIBILITY:
Inclusion Criteria for Providers:

* All providers that are part of Pathfinder Internal's supported clinic network in Burkina Faso, Tanzania, and Pakistan.

Exclusion Criteria for Providers:

* None

Inclusion Criteria for Clients:

* All clients aged 24 or under that visit a clinic that is enrolled in the study

Exclusion Criteria for Providers:

* Clients over 24
* Clients who do not visit the clinic for family planning services

Max Age: 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — This study is about family planning for women so we do not incldude men in the study
Enrollment: 233 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Whether client was able to receive services | 12 months after the intervention starts
  This is a measure of whether the client received family planning services on the day they came into the clinic. This will be measured from real clients using client exit surveys and using mystery clients.
Optimal Counseling | 12 months after the intervention starts
  This is a measure of whether the client was counseled on all methods that were good options for the client given her background and preferences. This will be coded as 1 if client was counseled on the full set of optimal family planning methods and zero if the client was not counseled on the full set of optimal family planning methods. This will be collected in the client exit survey and in by mystery clients.
Received modern method | 12 months after the intervention starts
  This is a measure of whether the client received a modern family planning method during her visit. This will be collected in the client exit survey only.
Perceived patient centeredness | 12 months after the intervention starts
  This is a composite scale (ranging from 0 to 1) that measures the extent to which the client perceived the her interaction with family provider as patient centered. The questions included in the scale will be chosen based on data driven factor analysis methods. Higher scores will indicate better patient centeredness. This will be collected in the client exit survey and in by mystery clients.

SECONDARY OUTCOMES:
Provider biased attitudes | 12 months after the intervention starts
  This is a composite scale (ranging from 0 to 1) that measures the extent to which providers have biased attitudes towards young, unmarried, and adolescent women. The questions included in the scale will be chosen based on data driven factor analysis methods. Higher scores will indicate better patient centeredness. This will be collected through a provider survey.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Wagner, Ph.D, Principal Investigator — RAND; Corrina Moucheraud, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- RAND, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected as part of the study and underlying results in publications will be de-identified and made public, with the exception of the content of in-depth interviews. IPD to be made available include data collected through provider surveys, mystery client visit debrief forms, and direct observations of client-provider interactions.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be made indefinitely available 6 months after publication.
Access Criteria: IPD will be made public, without any need for prior request.